CLINICAL TRIAL: NCT04818346
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose Ranging Study of the Efficacy and Safety of INCB054707 Followed by an Extension Period in Participants With Vitiligo
Brief Title: A Study to Evaluate the Efficacy and Safety of INCB054707 in Participants With Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB 54707-205
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Results first posted 2023-07-05 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: NonSegmental Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- INCB054707 Dose A followed by Dose C (Experimental): Participants will receive INCB054707 Dose A for 24 weeks (Period 1) followed by INCB054707 Dose C for 28 weeks (Period 2).
  Interventions: Drug: INCB054707
- INCB054707 Dose B (Experimental): Participants will receive INCB054707 Dose B for 52 weeks (Period 1 + Period 2).
  Interventions: Drug: INCB054707
- INCB054707 Dose C (Experimental): Participants will receive INCB054707 Dose C for 52 weeks (Period 1 + Period 2).
  Interventions: Drug: INCB054707
- Placebo followed by INCB054707 Dose C (Placebo Comparator): Participants will receive placebo for 24 weeks (Period 1) followed by INCB054707 Dose C for 28 weeks (Period 2).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INCB054707 — INCB054707 will be administered once daily
  Other Names: Povorcitinib
  Arms: INCB054707 Dose A followed by Dose C; INCB054707 Dose B; INCB054707 Dose C
Drug: Placebo — Placebo or INCB054707 will be administered once daily
  Arms: Placebo followed by INCB054707 Dose C

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of INCB054707 over a 24-week placebo-controlled double-blind treatment period, followed by a 28-week double-blind extension period in participants with nonsegmental vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of nonsegmental vitiligo.
* History of prior vitiligo treatment with a total duration of at least 3 months.
* Agreement to discontinue all agents and procedures used to treat vitiligo from screening through the final safety follow-up visit.
* Willingness to avoid pregnancy or fathering children
* Further inclusion criteria apply.

Exclusion Criteria:

* Other forms of vitiligo (eg, segmental) or other skin depigmentation disorders.
* Uncontrolled thyroid function at screening as determined by the investigator.
* Women who are pregnant (or who are considering pregnancy) or lactating.
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, Q-wave interval abnormalities, current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator.
* Have evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis.
* Participants known to be infected with HIV, Hepatitis B, or Hepatitis C.
* Laboratory values outside of the protocol-defined ranges.
* Further exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (23):
  - Investigative Site 010, Hoover, Alabama
  - Investigative Site 015, Gilbert, Arizona
  - Investigative Site 028, Scottsdale, Arizona
  - Investigative Site 006, Irvine, California
  - Investigative Site 009, Los Angeles, California
  - Investigative Site 018, Los Angeles, California
  - Investigative Site 017, Sacramento, California
  - Investigative Site 032, Orange Park, Florida
  - Investigative Site 005, Tampa, Florida
  - Investigative Site 022, Tampa, Florida
  - Investigative Site 011, West Palm Beach, Florida
  - Investigative Site 024, Covington, Louisiana
  - Investigative Site 002, Brighton, Massachusetts
  - Investigative Site 023, Saint Paul, Minnesota
  - Investigative Site 027, Verona, New Jersey
  - Investigative Site 003, Columbus, Ohio
  - Investigative Site 007, Norman, Oklahoma
  - Investigative Site 001, Portland, Oregon
  - Investigative Site 021, Plymouth Meeting, Pennsylvania
  - Investigative Site 004, Murfreesboro, Tennessee
  - Investigative Site 033, Dallas, Texas
  - Investigative Site 012, San Antonio, Texas
  - Investigative Site 030, Spokane, Washington
- Canada (8):
  - Investigative Site 020, Winnipeg, Manitoba
  - Investigative Site 014, Etobicoke, Ontario
  - Investigative Site 034, London, Ontario
  - Investigative Site 025, Mississauga, Ontario
  - Investigative Site 026, North YORK, Ontario
  - Investigative Site 031, Oakville, Ontario
  - Investigative Site 008, Peterborough, Ontario
  - Investigative Site 029, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in 28 sites in Canada and the United States.
Groups:
- Placebo: Participants received matching placebo QD for 24 weeks (placebo-controlled period). Participants who completed the Week 24 visit received oral povorcitinib 75 mg QD for an additional 28 weeks (double-blind extension period).
- Povorcitinib 15 mg: Participants received oral povorcitinib 15 milligrams (mg) once daily (QD) for 24 weeks (placebo-controlled period). Participants who completed the Week 24 visit received oral povorcitinib 75 mg QD for 28 weeks (double-blind extension period).
- Povorcitinib 45 mg: Participants received oral povorcitinib 45 mg QD for 24 weeks (placebo-controlled period). Participants who completed the Week 24 visit received oral povorcitinib 45 mg QD for an additional 28 weeks (double-blind extension period).
- Povorcitinib 75 mg: Participants received oral povorcitinib 75 mg QD for 24 weeks (placebo-controlled period). Participants who completed the Week 24 visit received oral povorcitinib 75 mg QD for an additional 28 weeks (double-blind extension period.
Period: 24-Week Placebo-controlled Period
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Started | 43 | 43 | 43 | 42
Completed | 35 | 38 | 32 | 34
Not Completed | 8 | 5 | 11 | 8
Not completed — Adverse Event | 1 | 2 | 0 | 3
Not completed — Lost to Follow-up | 3 | 2 | 3 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 6 | 2
Not completed — Subject Terminated by Sponsor | 1 | 0 | 0 | 0
Not completed — Latent Tuberculosis; Unable to Provide Proof of Treatment | 1 | 0 | 0 | 0
Not completed — Use of Prohibited Concomitant Medication | 0 | 0 | 1 | 0
Not completed — Ineligible to Be Included in the Study Due to Abnormal Coagulation Profile | 0 | 0 | 0 | 1
Period: 28-Week Double-blind Extension Period
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Started | 35 | 37 | 32 | 34
Completed | 33 | 30 | 26 | 28
Not Completed | 2 | 7 | 6 | 6
Not completed — Adverse Event | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 4 | 3
Not completed — Non-compliance | 0 | 1 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 1 | 0 | 0
Not completed — Scheduling Conflicts | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg | Total
Number analyzed (Participants) | 43 | 43 | 43 | 42 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (12.92) | 45.9 (11.56) | 50.2 (11.61) | 50.5 (11.69) | 48.8 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 21 | 19 | 93
  Male | 19 | 14 | 22 | 23 | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 34 | 32 | 38 | 28 | 132
  Black/African-American | 2 | 3 | 1 | 3 | 9
  Asian | 2 | 4 | 0 | 7 | 13
  Mexican American | 1 | 0 | 0 | 0 | 1
  African-European | 1 | 0 | 0 | 0 | 1
  Middle Eastern | 0 | 1 | 1 | 0 | 2
  Columbian | 0 | 0 | 0 | 1 | 1
  Captured as Hispanic in Database | 0 | 0 | 0 | 2 | 2
  Mixed | 0 | 1 | 0 | 0 | 1
  Mexican | 0 | 0 | 1 | 0 | 1
  East Indian | 1 | 0 | 0 | 0 | 1
  Did Not Identify with Options Provided | 0 | 1 | 0 | 0 | 1
  White and Asian-Non-Japanese | 0 | 0 | 1 | 0 | 1
  South African | 0 | 1 | 0 | 0 | 1
  White/Black | 1 | 0 | 0 | 0 | 1
  South American | 0 | 0 | 0 | 1 | 1
  Egyptian | 0 | 0 | 1 | 0 | 1
  Captured as Hispanic/Latino in Database | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 11 | 7 | 32
  Not Hispanic or Latino | 35 | 36 | 32 | 34 | 137
  Not Reported | 0 | 0 | 0 | 1 | 1
  Bangladeshi | 0 | 1 | 0 | 0 | 1
Total Vitiligo Area Scoring Index (T-VASI) [Mean (Standard Deviation); unit: scores on a scale] — The T-VASI was calculated based on values from 6 body regions (possible range: 0-100; higher values=worse outcome). The percentage of vitiligo involvement was estimated in hand units (% body surface area [BSA]; investigator assessed), based on the participant's hand size. The degree of depigmentation for each body site was determined and estimated to the nearest percentage: 0%, 10%, 25%, 50%, 75%, 90%, or 100%. The T-VASI was derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each body site and summing the values of all body sites.
  scores on a scale | 28.31 (21.481) | 27.13 (20.085) | 23.64 (19.758) | 22.65 (14.244) | 25.45 (19.094)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Vitiligo Area Scoring Index (T-VASI) at Week 24
Description: The T-VASI was calculated based on values from the whole body, which was split into 6 separate and mutually exclusive regions (possible range: 0-100; higher values=worse outcome). The percentage of vitiligo involvement was estimated in hand units (% body surface area [BSA]; investigator assessed), based on the participant's hand size. The degree of depigmentation for each body site was determined and estimated to the nearest percentage: 0%, 10%, 25%, 50%, 75%, 90%, or 100%. The T-VASI was derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each body site and summing the values of all body sites. Percent change was calculated as ([post-Baseline value minus the Baseline value] / Baseline value) x 100.
Time Frame: Baseline; Week 24
Population: Intent-to-Treat Population: all randomized participants. Treatment groups for this population were defined according to the treatment assignment at randomization. Mixed-effect model for repeated measures (MMRM) model: (percent change from Baseline = treatment + stratification factor [T-BSA involvement 8%-20%/>20%] + visit + treatment*visit + Baseline measurement + Baseline measurement*visit). Only participants with available data were analyzed.
Measure: Geometric Least Squares Mean (Standard Error); unit: percent change
Groups:
- Povorcitinib 75 mg: Participants received oral povorcitinib 75 mg QD for 24 weeks (placebo-controlled period). Participants who completed the Week 24 visit received oral povorcitinib 75 mg QD for an additional 28 weeks (double-blind extension period).
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 33 | 38 | 33 | 36
percent change | 2.29 (4.81) | -19.12 (4.56) | -17.78 (4.87) | -15.73 (4.74)
Statistical Analysis 1: Comparison: Placebo vs Povorcitinib 15 mg; Test type: Superiority; p = 0.0015, Mixed Model Repeated Measures (MMRM); Least squares mean difference = -21.41, 95% CI 2-sided [-34.49 to -8.32], Standard Error of Mean 6.62
Statistical Analysis 2: Comparison: Placebo vs Povorcitinib 45 mg; Test type: Superiority; p = 0.0040, MMRM; Least squares mean difference = -20.07, 95% CI 2-sided [-33.63 to -6.51], Standard Error of Mean 6.86
Statistical Analysis 3: Comparison: Placebo vs Povorcitinib 75 mg; Test type: Superiority; p = 0.0086, MMRM; Least squares mean difference = -18.02, 95% CI 2-sided [-31.40 to -4.64], Standard Error of Mean 6.77

2. Secondary Outcome: Percentage of Participants Achieving T-VASI50 at Week 24
Description: T-VASI50 was defined as a 50% or greater reduction from Baseline in T-VASI. The T-VASI was calculated based on values from the whole body, which was split into 6 separate and mutually exclusive body regions (possible range: 0-100; higher values=worse outcome). The percentage of vitiligo involvement was estimated in hand units (% body surface area [BSA]; investigator assessed), based on the participant's hand size. The degree of depigmentation for each body site was determined and estimated to the nearest percentage: 0%, 10%, 25%, 50%, 75%, 90%, or 100%. The T-VASI was derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each body site and summing the values of all body sites.
Time Frame: Baseline; Week 24
Population: Intent-to-Treat Population. The 95% confidence interval was based on the Clopper-Pearson exact method. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 43 | 43 | 43 | 42
percentage of participants | 2.3 [0.1 to 12.3] | 9.3 [2.6 to 22.1] | 11.6 [3.9 to 25.1] | 4.8 [0.6 to 16.2]
Statistical Analysis 1: Comparison: Placebo vs Povorcitinib 15 mg; Test type: Superiority; p = 0.3574, Wald test; Odds Ratio (OR) = 4.3, 95% CI 2-sided [0.398 to 220.998] — Logistic regression: (response at Week 24 = treatment + stratification factor [T-BSA involvement 8%-20%/>20%])
Statistical Analysis 2: Comparison: Placebo vs Povorcitinib 45 mg; Test type: Superiority; p = 0.1992, Wald test; Odds Ratio (OR) = 5.5, 95% CI 2-sided [0.573 to 273.479] — Logistic regression: (response at Week 24 = treatment + stratification factor [T-BSA involvement 8%-20%/>20%])
Statistical Analysis 3: Comparison: Placebo vs Povorcitinib 75 mg; Test type: Superiority; p = 0.9913, Wald test; Odds Ratio (OR) = 2.1, 95% CI 2-sided [0.103 to 126.386] — Logistic regression: (response at Week 24 = treatment + stratification factor [T-BSA involvement 8%-20%/>20%])

3. Secondary Outcome: Placebo-controlled Period: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of the study drug. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until the end of the safety follow-up period.
Time Frame: up to Week 24
Population: Safety Population: all participants who received at least 1 dose of study drug. Treatment groups for this population were to have been determined according to the actual treatment the participant received on Day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 42 | 43 | 41 | 42
Participants | 24 | 29 | 30 | 35

4. Secondary Outcome: Extension Period: Number of Participants With Any TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of the study drug. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug until the end of the safety follow-up period.
Time Frame: from Week 25 up to Week 76
Population: Extension Evaluable Population: all participants who received at least 1 dose of povorcitinib during the double-blind extension period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
Number analyzed (Participants) | 35 | 37 | 32 | 34
Participants | 27 | 28 | 21 | 31

ADVERSE EVENTS:
Time Frame: up to Week 76
Description: Treatment-emergent adverse events (TEAEs) occurring in the placebo-controlled period have been reported for members of the Safety Population (all participants who received at least 1 dose of povorcitinib or placebo during the placebo-controlled period). TEAEs occurring in the double-blind extension period have been reported for members of the Extension Evaluable Population (participants who received at least 1 dose of povorcitinib during the double-blind extension period).
Groups:
- Povorcitinib 75 mg: Participants received placebo, oral povorcitinib 15 mg QD, or oral povorcitinib 75 mg QD for 24 weeks (placebo-controlled period). Participants who completed the Week 24 visit received oral povorcitinib 75 mg QD for an additional 28 weeks (double-blind extension period).
Arm/Group | Placebo | Povorcitinib 15 mg | Povorcitinib 45 mg | Povorcitinib 75 mg
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/43 | 0/41 | 0/114
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/43 | 1/41 | 1/114
Other Adverse Events (participants affected / at risk) | 19/42 | 22/43 | 24/41 | 69/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | Povorcitinib 15 mg (N=43) | Povorcitinib 45 mg (N=41) | Povorcitinib 75 mg (N=114)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | Povorcitinib 15 mg (N=43) | Povorcitinib 45 mg (N=41) | Povorcitinib 75 mg (N=114)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 22 (28)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 4 (5) | 4 (4)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 3 (3) | 4 (6) | 21 (25)
COVID-19 (Infections and infestations) | 5 (5) | 8 (8) | 13 (14) | 31 (31)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Fatigue (General disorders) | 2 (2) | 3 (3) | 3 (3) | 7 (7)
Headache (Nervous system disorders) | 5 (5) | 7 (9) | 1 (1) | 9 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (3) | 9 (11)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2) | 6 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 6 (7) | 6 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 4 (5) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT04818346/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT04818346/SAP_001.pdf